CLINICAL TRIAL: NCT03767699
Title: Medical Nutrition Therapy Program and Eating Behavior Questionnaires on Gestational Weight Gain in Mexican Women With Diabetes
Brief Title: Medical Nutrition Therapy Program and Eating Behavior Questionnaires on Gestational Weight Gain
Status: Completed | Type: Observational
Sponsor: Hugo Mendieta Zeron (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Sponsor-Investigator, Hugo Mendieta Zeron, Chief of the Research Department, Materno-Perinatal Hospital of the State of Mexico
Organization: Materno-Perinatal Hospital of the State of Mexico (Other)
Other Study IDs: 2013-12-239; D43TW009135 (NIH)
Record Dates: First submitted 2018-12-04; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Gestational Weight Gain
Keywords: Medical nutrition therapy; Eating behavior; Type 2 diabetes mellitus; Gestational Diabetes
MeSH Terms: conditions — Gestational Weight Gain; Feeding Behavior; Diabetes Mellitus, Type 2; Diabetes, Gestational | interventions — Nutrition Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Medical Nutrition Therapy — MNT was offered every 2-4 weeks to all pregnant women with T2DM and GDM. Women. MNT is offered as a mandatory part of their prenatal visit and/or hospital stay. The MNT provides an individual food plan with the following recommendations: total calories should be calculated as 30 kcal/kg based on pregestational BMI for an ideal weight. Of the total energy intake 40-45% is provided by carbohydrates, a maximum of 40% is provided by lipids and the remaining percentage by proteins providing moderate-to-low glycemic index foods and fiber consumption, glucose self-monitoring, participating in 15-30 min of daily physical activity after prior authorization of the treating physician, and meeting the minimal energy requirements of pregnancy (never < 1,500 kcal).

SUMMARY:
Type 2 Diabetes Mellitus (T2DM) and Gestational Diabetes Mellitus (GDM) create complications during pregnancy, particularly in women with gestational weight gain (GWG) that falls over the recommended limit. On the other hand Medical nutrition therapy (MNT) has been shown to reduce some complications in women with T2DM and GDM. The aim of this project was to assess the association of MNT consultations and eating behavior with GWG in Mexican women with T2DM and GDM.

DETAILED DESCRIPTION:
This cross-sectional study conducted at from 2013 to 2014. Fifty seven patients with T2DM or GDM were invited to participate. The dependent variable was GWG and the main independent variables were MNT and eating behaviors. Data were obtained from medical records or interviews. Multiple linear regression models were used to assess associations.

ELIGIBILITY:
Inclusion Criteria:

* Women who had given birth and with known T2DM.
* Women who had given birth and with GDM diagnosed during pregnancy.

Exclusion Criteria:

* Women with multiple pregnancies.
* Women with type 1 diabetes mellitus.
* Women with glucose intolerance.
* Women with chronic diseases.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women with T2DM or GDM who received as a routine management the Medical Nutrition Therapy. The characteristics of the pregnant women usually attended at the Maternal-Perinatal Hospital "Mónica Pretelini Sáenz" are: low socioecomic status and education, they all receive free medical attention.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Gestational Weight Gain | Nine months
  Weight (kg) was measured using a weight scale (SECA 711). GWG was calculated by subtracting the prepregnancy weight from the weight at the end of the third trimester (kg). Recommended GWG was based on U.S. Institute of Medicine guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Garduño Alanís, PhD., Study Chair — Independent researcher.
Locations (1):
- Materno-Perinatal Hospital "Mónica Pretelini", Toluca, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Information will be available upon request.

REFERENCES:
- [Background] Horosz E, Bomba-Opon DA, Szymanska M, Wielgos M. Maternal weight gain in women with gestational diabetes mellitus. J Perinat Med. 2013 Sep 1;41(5):523-8. doi: 10.1515/jpm-2012-0254. PMID 23492551
- [Background] Perichart-Perera O, Balas-Nakash M, Parra-Covarrubias A, Rodriguez-Cano A, Ramirez-Torres A, Ortega-Gonzalez C, Vadillo-Ortega F. A medical nutrition therapy program improves perinatal outcomes in Mexican pregnant women with gestational diabetes and type 2 diabetes mellitus. Diabetes Educ. 2009 Nov-Dec;35(6):1004-13. doi: 10.1177/0145721709343125. Epub 2009 Aug 20. PMID 19696205
- [Background] Balas-Nakash M, Rodriguez-Cano A, Munoz-Manrique C, Vasquez-Pena P, Perichart-Perera O. [Adherence to a medical nutrition therapy program in pregnant women with diabetes, measured by three methods, and its association with glycemic control]. Rev Invest Clin. 2010 May-Jun;62(3):235-43. Spanish. PMID 20815129
- [Background] Jaakkola J, Hakala P, Isolauri E, Poussa T, Laitinen K. Eating behavior influences diet, weight, and central obesity in women after pregnancy. Nutrition. 2013 Oct;29(10):1209-13. doi: 10.1016/j.nut.2013.03.008. Epub 2013 Jun 22. PMID 23800568
- [Derived] Garduno-Alanis A, Torres-Mejia G, Nava-Diaz P, Herrera-Villalobos J, Diaz-Arizmendi D, Mendieta-Zeron H. Association between a medical nutrition therapy program and eating behavior with gestational weight gain in women with diabetes. J Matern Fetal Neonatal Med. 2020 Dec;33(24):4049-4054. doi: 10.1080/14767058.2019.1594764. Epub 2019 Mar 28. PMID 30880554